CLINICAL TRIAL: NCT00965263
Title: Tests of a Therapeutic Cocaine Vaccine
Brief Title: Therapeutic Cocaine Vaccine: Human Laboratory Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #3980; NIDA 1U19DA10946
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-09

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; immunotherapy; vaccination; antibody; addiction; dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose Vaccine (Experimental): All participants were vaccinated four times: in week 1, 3, 5, and 9. Dose: 82ul
  Interventions: Biological: Cocaine vaccine (TA-CD)
- High Dose Vaccine (Experimental): All participants were vaccinated four times: in week 1, 3, 5, and 9. Dose: 360ul
  Interventions: Biological: Cocaine vaccine (TA-CD)

INTERVENTIONS:
Biological: Cocaine vaccine (TA-CD) — TA-CD (82,360 μg; IM) were administered at weeks 1, 3, 5 and 9.

SUMMARY:
Clinical data demonstrate that a cocaine vaccine (TA-CD: Celtic Pharmaceutical) produces selective anti-cocaine antibodies, yet the impact of these antibodies on cocaine's direct effects is unknown. The objective of this human laboratory study was to measure the relationship between antibody titers and the effects of smoked cocaine on ratings of intoxication, craving and cardiovascular effects.

Cocaine-dependent volunteers not seeking drug treatment spend 2 nights per week for 13 weeks inpatient where the effects of cocaine (0, 25, 50 mg) are determined prior to vaccination and at weekly intervals thereafter. Vaccinations occur at weeks 1, 3, 5 and 9.

DETAILED DESCRIPTION:
I do not desire to provide a more extensive description.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV criteria for current cocaine dependence. The volunteer may meet criteria for other substance abuse, but not dependence (other than nicotine).
2. Primary route of cocaine administration is smoking.
3. Age 21-45.
4. Females must be surgically sterilized or post- menopausal
5. Able to give informed consent, and comply with study procedures.

Exclusion Criteria:

1. Dependence on substances other than cocaine or nicotine.
2. Judged to be noncompliant with study protocol.
3. History of autoimmune disease, immune deficiency or hypersensitivity to other vaccines. An HIV test must be negative.
4. Currently uses drugs intravenously
5. Currently taking any psychotropic medication
6. Laboratory tests that are clinically unacceptable to the study physician (BP > 140/90; BUN, creatinine, LFTs > 1.5 ULN; hematocrit < 34 for women, < 36 for men)
7. Blood or blood products given in the three months prior to vaccination
8. Other vaccines, including flu vaccine, given within 30 days of screening.
9. Ongoing active infection
10. Currently taking immunosuppressives -

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — Columbia University
Locations (1):
- New York-Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Derived] Haney M, Gunderson EW, Jiang H, Collins ED, Foltin RW. Cocaine-specific antibodies blunt the subjective effects of smoked cocaine in humans. Biol Psychiatry. 2010 Jan 1;67(1):59-65. doi: 10.1016/j.biopsych.2009.08.031. PMID 19846066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cocaine-dependent research volunteers who were explicitly not interested in treatment for their cocaine use signed a consent form approved by NYSPI IRB, which described the procedures and outlined the possible risks, including administration of an experimental vaccine and smoked cocaine.
Groups:
- Low Dose Vaccine: All participants were vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (82 μg; IM) were administered at weeks 1, 3, 5 and 9.
- High Dose Vaccine: All participants were vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (360 μg; IM) were administered at weeks 1, 3, 5 and 9.
Period: Overall Study
Arm/Group | Low Dose Vaccine | High Dose Vaccine
Started | 6 | 9
Completed | 4 | 6
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Family emergency | 0 | 1
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Overall, 10 volunteers participated in this study.
Groups:
- Low Dose Vaccine (82μg): All participants were vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (82 μg; IM) were administered at weeks 1, 3, 5 and 9.
- High Dose Vaccine (360μg): All participants were vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (360 μg; IM) were administered at weeks 1, 3, 5 and 9.
- Total: Total of all reporting groups
Arm/Group | Low Dose Vaccine (82μg) | High Dose Vaccine (360μg) | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (1.8) | 39 (1.9) | 39 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 1 | 2 | 3
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Intoxication
Description: Visual Analogue Scale ratings (0-100mm) of the Good Drug Effect cluster ("Good Drug Effect," "High," "Stimulated") over 13 weeks as a function of cocaine dose (25mg or 50mg). Participants (n=10) were evenly divided into High Antibody (AB) and Low Antibody (AB) groups based on their peak antibody levels at Week 13. Higher numbers indicate more agreement with the statements.
Time Frame: 13 weeks
Population: Peak plasma antibody levels were highly variable. Thus, participants (n=10) were evenly divided into High Antibody (AB) and Low Antibody (AB) groups for analysis, based on their peak antibody levels at Week 13, rather than by the dose of vaccine received.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Week 1 Low Antibody; Week 3 Low Antibody; Week 5 Low Antibody; Week 7 Low Antibody; Week 9 Low Antibody; Week 11 Low Antibody; Week 13 Low Antibody; Week 1 High Antibody; Week 3 High Antibody; Week 5 High Antibody; Week 7 High Antibody; Week 9 High Antibody; Week 11 High Antibody; Week 13 High Antibody: Participants were evenly divided into low antibody and high antibody groups based on their peak antibody levels at week 13.
Arm/Group | Week 1 Low Antibody | Week 3 Low Antibody | Week 5 Low Antibody | Week 7 Low Antibody | Week 9 Low Antibody | Week 11 Low Antibody | Week 13 Low Antibody | Week 1 High Antibody | Week 3 High Antibody | Week 5 High Antibody | Week 7 High Antibody | Week 9 High Antibody | Week 11 High Antibody | Week 13 High Antibody
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
units on a scale
  Good Drug Effect of 25 mg cocaine | 59 (9) | 51 (8) | 45 (9) | 44 (8) | 42 (8) | 38 (8) | 40 (7) | 58 (8) | 32 (8) | 29 (0) | 23 (4) | 29 (3) | 19 (3) | 10 (2)
  Good Drug Effect of 50 mg cocaine | 83 (4) | 68 (8) | 61 (7) | 58 (8) | 58 (8) | 50 (10) | 60 (8) | 62 (8) | 50 (8) | 48 (4) | 48 (8) | 42 (6) | 48 (5) | 25 (5)

2. Secondary Outcome: Cocaine Cardiovascular Effects
Description: Heart rate levels in Week 3 and Week 13 as a function of cocaine dose in High and Low antibody groups. Participants (n=10) were evenly divided into High Antibody (AB) and Low Antibody (AB) groups based on their peak antibody levels at Week 13. Higher numbers indicate higher heart rates.
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: BPM
Groups:
- Low Antibody/0mg Cocaine: Low Antibody/0mg Cocaine.
- Low Antibody/25mg Cocaine: Low Antibody/25mg Cocaine.
- Low Antibody/50mg Cocaine: Low Antibody/50mg Cocaine.
- High Antibody/0mg Cocaine: High Antibody/0mg Cocaine.
- High Antibody/25mg Cocaine: High Antibody/25mg Cocaine.
- High Antibody/50mg Cocaine: High Antibody/50mg Cocaine.
Arm/Group | Low Antibody/0mg Cocaine | Low Antibody/25mg Cocaine | Low Antibody/50mg Cocaine | High Antibody/0mg Cocaine | High Antibody/25mg Cocaine | High Antibody/50mg Cocaine
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
BPM
  Week 3 | 75 (3) | 82 (2) | 92 (1) | 79 (1.5) | 98 (3) | 109 (4)
  Week 13 | 76 (2) | 99 (2) | 102 (2) | 82 (2) | 101 (5) | 122 (6)

3. Secondary Outcome: Plasma Cocaine
Description: Plasma cocaine levels in Week 3 and Week 13 as a function of cocaine dose in High and Low AB groups. Participants (n=10) were evenly divided into High Antibody (AB) and Low Antibody (AB) groups based on their peak antibody levels at Week 13. Higher numbers indicate higher plasma levels of cocaine.
Time Frame: 13 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Low Antibody/0mg Cocaine | Low Antibody/25mg Cocaine | Low Antibody/50mg Cocaine | High Antibody/0mg Cocaine | High Antibody/25mg Cocaine | High Antibody/50mg Cocaine
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
ng/mL
  Week 3 | 5 (0.2) | 125 (8) | 160 (10) | 20 (2) | 145 (20) | 260 (40)
  Week 13 | 25 (2) | 110 (5) | 200 (20) | 25 (2) | 175 (10) | 325 (50)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Low Dose Vaccine: Each of four participants was vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (82 μg; IM) were administered at weeks 1, 3, 5 and 9.
- High Dose Vaccine: Each of six participants was vaccinated four times: in week 1, 3, 5, and 9.
  Cocaine vaccine (TA-CD): TA-CD (360 μg; IM) were administered at weeks 1, 3, 5 and 9.
Arm/Group | Low Dose Vaccine | High Dose Vaccine
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

LIMITATIONS AND CAVEATS:
There was no placebo TA-CD condition, due to the substantial study demands.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes